CLINICAL TRIAL: NCT06629714
Title: Cohort Studies of Impact of Pretreatment Emotional on Survival and the Predictive Role of Peripheral Blood Metabolic and Inflammatory Markers in Immunotherapy Response Among Treatment-Naïve, Advanced and Inoperable Gastroesophageal and Non-Small-Cell Lung Cancer Patients
Brief Title: Impact of Pretreatment Emotional Distress on Survival and the Predictive Role of Peripheral Biomarkers in Immunotherapy Response Among Gastroesophageal and Lung Cancer Patients
Status: Completed | Type: Observational
Sponsor: Anhui Medical University (Other)
Responsible Party: Principal Investigator, Huaidong Cheng, Professor, Anhui Medical University
Other Study IDs: 83242393
Record Dates: First submitted 2024-10-04; First posted 2024-10-08 (Actual); Last update posted 2026-01-13 (Actual); Status verified 2026-01

CONDITIONS: Non Small Cell Lung Cancer; Immune Checkpoint Inhibitors; Inflammation; Cancer, Treatment-Related; Emotional Distress; Gastroesophageal Cancer (GC); Biomarkers / Blood; Progression-free Survival, PFS
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Inflammation; Neoplasms, Second Primary

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Cohort 1: Treatment-naïve, advanced and inoperable GEC patients receiving first-line ICIs: For treatment-naïve, advanced and inoperable Esophageal Cancer or Gastric Cancer or Gastroesophageal junction (GEJ) Cancer patients who have received immune checkpoint inhibitors as first-line therapy.
  Interventions: Other: Exposure: emotional distress status
- Cohort 2: Treatment-naïve, advanced and inoperable NSCLC patients receiving first-line ICIs.: For treatment-naïve, advanced and inoperable Non-Small-Cell Lung Cancer patients who have received immune checkpoint inhibitors as first-line therapy.
  Interventions: Other: Exposure: emotional distress status

INTERVENTIONS:
Other: Exposure: emotional distress status — The assessment of depressive and anxiety symptoms was conducted using Patient Health Questionnaire-9 (PHQ-9) and Generalized Anxiety Disorder Assessment 7 (GAD-7). Patients with a sum score of PHQ-9 and GAD-7 ≥ 10 were categorized as the stressed group.

SUMMARY:
This is the prospective, observational cohort study to explore the impact of pretreatment emotional distress on survival and the predictive role of peripheral blood metabolic and inflammatory markers in immunotherapy response among treatment-naïve, advanced and inoperable Gastroesophageal Cancer (GEC) and non-small-cell lung cancer (NSCLC).

DETAILED DESCRIPTION:
This is the prospective, observational cohort study to explore the impact of pretreatment emotional distress on survival and the predictive role of peripheral blood metabolic and inflammatory markers in immunotherapy response among treatment-naïve, advanced and inoperable Gastroesophageal Cancer (GEC) and Non-Small-Cell Lung Cancer (NSCLC). Eligible patients were administered first-line treatment with either immune checkpoint inhibitor or a combination of immunotherapy and chemotherapy upon enrollment. This study will have 2 cohorts:

* Cohort 1: A prospective, observational cohort study to explore the impact of pretreatment emotional distress on survival and the predictive role of peripheral blood metabolic and inflammatory markers in immunotherapy response among treatment-naïve, advanced and inoperable GEC patients.
* Cohort 2: A prospective, observational cohort study to explore the impact of pretreatment emotional distress on survival and the predictive role of peripheral blood metabolic and inflammatory markers in immunotherapy response among treatment-naïve, advanced and inoperable NSCLC patients.

ELIGIBILITY:
Cohort 1 & 2

Inclusion Criteria:

* Meet the diagnostic criteria for cancer (including esophageal, gastric, GEJ or NSCLC) through clinical, pathological, and imaging examinations;
* Karnofsky Performance Status (KPS) score should be equal to or greater than 80 points;
* Unresectable locally advanced or metastatic;
* Systematic treatments naive ( e. g., chemotherapy, anti-angiogenic drugs, targeted drugs, and immunotherapy);
* Presence of at least one measurable lesion according to the Response Evaluation Criteria in Advanced Solid Tumors version 1.1 (RECIST v1.1);
* Receiving PD-1/PD-L1 inhibitors monotherapy or combination with chemotherapy;
* Informed and agreed to participate in the study;
* Required to complete the questionnaire independently or with assistance from others if needed;
* Legal age, 18 years or older.

Exclusion Criteria:

* Oncogene-driver positive;
* Combined with other malignant tumors in the past 3 years;
* Concurrent acute or chronic psychiatric disorders;
* Current receiving anti-depressive or anti-anxiety therapy or other psychotropic drugs;
* Previous treatment with other clinical drug trials;
* Patients with symptomatic brain metastasis;
* Severe intellectual disabilities or other communication difficulties that hindered normal interaction.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Cohort 1 comprises patients diagnosed with treatment-naïve, advanced and inoperable Gastroesophageal Cancer (GEC), encompassing those with esophageal cancer, gastric cancer, and gastroesophageal junction cancer who are undergoing first-line ICI therapy. Cohort 2 consists of patients with treatment-naïve, advanced and inoperable Non-Small Cell Lung Cancer (NSCLC) receiving first-line ICI therapy.
Sampling Method: Probability Sample
Enrollment: 196 (Actual)
Dates: Start 2020-10-16 (Actual); Primary Completion 2025-04-20 (Actual); Study Completion 2025-04-20 (Actual)

PRIMARY OUTCOMES:
Cohort 1 & 2: Progression-free survival (PFS) | 4 year
  Time from the beginning of first-line immunotherapy to the first progression (PD) or death in patients

SECONDARY OUTCOMES:
Value of Neutrophils to lymphocytes ratio (NLR) | 0 day, 6 weeks
  NLR is an inflammatory marker, which is the ratio of neutrophils to lymphocytes. The higher the value is, the higher the inflammatory level may be. The information has been extracted from the medical record and evaluated longitudinally.
Value of Platelet-lymphocyte ratio (PLR) | 0 day, 6 weeks
  PLR is an inflammatory marker, a ratio of platelets to lymphocytes. A higher value of it indicates a higher level of inflammation in the body. The information has been extracted from the medical record and evaluated longitudinally.
Value of Monocyte-lymphocyte ratio (MLR) | 0 day, 6 weeks
  MLR is an inflammatory indicator, which is the ratio of macrophages and lymphocytes. The higher the value is, the higher the inflammatory level in the body is. The information has been extracted from the medical record and evaluated longitudinally.
Value of Systemic immune inflammation index (SII) | 0 day, 6 weeks
  SII is an inflammatory indicator, which is calculated as follows: SII= (neutrophil × platelet)/lymphocytes. A higher value indicates an elevated level of inflammation within the body. The information has been extracted from the medical record and evaluated longitudinally.
Value of Pan-immune inflammation value (PIV) | 0 day, 6 weeks
  PIV is an inflammatory indicator, which is equal to neutrophils × monocytes × platelets/lymphocytes. The higher the value is, the higher the inflammatory level in the body is. The information has been extracted from the medical record and evaluated longitudinally.
Value of eosinophil fraction | 0 day, 6 weeks
  The eosinophil fraction is a potential inflammation and tumor prognostic indicator, which equals the ratio of eosinophil absolute value to the total white blood cell count. The higher the value of this fraction, the better the tumor prognosis may be. The information has been extracted from the medical record and evaluated longitudinally.
Value of prognostic nutritional index (PNI) | 0 day, 6 weeks
  PNI is a potential inflammation and tumor prognostic indicator, which is equal to albumin level (g/L) + 5 × absolute value of lymphocyte counts. The higher the value of this index, the better the tumor prognosis may be. The information has been extracted from the medical record and evaluated longitudinally.
Value of Blood glucose | 0 day, 6 weeks
  Blood glucose is an indicator of metabolism in the body. The information has been extracted from the medical record and evaluated longitudinally.
Value of Triglycerides | 0 day, 6 weeks
  Triglycerides is an indicator of metabolism in the body. The information has been extracted from the medical record and evaluated longitudinally.
Value of Total cholesterol | 0 day, 6 weeks
  Total cholesterol is an indicator of metabolism in the body. The information has been extracted from the medical record and evaluated longitudinally.
Value of Albumin | 0 day, 6 weeks
  Albumin is an indicator of metabolism in the body. The information has been extracted from the medical record and evaluated longitudinally.
Disease Control Rate (DCR) | 1 year
  DCR refers to the proportion of patients with tumor treated with a certain treatment who have tumor shrinkage or stable disease, and this state can be maintained for a certain period of time, including the proportion of Complete Response (CR), Partial Response (PR) and Stable Disease (SD).

OTHER OUTCOMES:
Prognostic models for immunotherapy | 0 day, 6 weeks
  Tumor biomarkers, such as CEA, CA19-9, CA72-4, NSE, SCC, and the above-mentioned metabolic and inflammatory markers in peripheral blood were collected at baseline and after two cycles of treatment (6 weeks). The scores of PHQ-9 and GAD-7 questionnaires were also collected. The variables were screened to establish an optimal prognostic model.

CONTACTS AND LOCATIONS:
Locations (1):
- Second Affiliated Hospital of Anhui Medical University, Hefei, Anhui, China

IPD SHARING:
Plan to Share IPD: No